CLINICAL TRIAL: NCT06504797
Title: The Effect of Automatic Massage Applied to Healthcare Workers on Pain, Fatigue and Psychological Well-being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Emine Yıldırım, Assistant Professor, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2345
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Massage; Pain, Back
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- massage group (Experimental): massage application
  Interventions: Device: automatic massage

INTERVENTIONS:
Device: automatic massage — automatic massage

SUMMARY:
To determine the effect of automatic massage applied to healthcare workers on pain, fatigue and psychological well-being. This research is planned as a pretest-posttest type study. It will be held in the Osmaniye State Hospital maternity ward. The application will be applied by one person in the rest room. Data will be collected using the Introductory Information Form, Psychological Well-Being Scale, Perceived Stress Scale (ASÖ/PSÖ-14), State-Trait Anxiety Inventory (STAI), and Piper Fatigue Scale.

ELIGIBILITY:
Inclusion Criteria:

* Working in the delivery room

Exclusion Criteria:

* Being receiving psychiatric treatment (Pharmacotherapy or psychotherapy),
* having a wound on the waist and back that prevents the application.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2024-07-26 (Estimated); Study Completion 2024-08-02 (Estimated)

PRIMARY OUTCOMES:
pain perception | 1 week
  pain scale